CLINICAL TRIAL: NCT06088264
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Pharmacokinetics, Metabolism, and Excretion of [14C] BMS-986322 in Healthy Adult Male Participants
Brief Title: A Study to Evaluate the Drug Levels, Metabolism, and Removal of BMS-986322 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM032-1018
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Healthy Male Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of BMS-986322 (Experimental)
  Interventions: Drug: BMS-986322

INTERVENTIONS:
Drug: BMS-986322 — Specified dose on specified days.

SUMMARY:
The purpose of this study is to evaluate the drug levels, metabolism, and removal of BMS-986322 in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index of 18.0 to 32.0 kg/m2, inclusive.
* Participants will be required to always use a latex or other synthetic condom with spermicide during any sexual activity
* Participants must refrain from donating sperm during the entire study and for at least 90 days from dose of study drug.

Exclusion Criteria:

* Participant must not have had any clinically significant diagnostic or therapeutic radiation exposure within the previous 12 months prior to admission to the clinic.
* Participant must not be currently employed in a job requiring radiation exposure monitoring.
* Participant must not have had any major surgery within 4 weeks of study drug administration that could impact upon the absorption of study drug

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed in plasma/whole blood concentration (Cmax) | Up to day 17
Area under the plasma/whole blood concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to day 17
Area under the plasma/whole blood concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to day 17
Time of maximum observed in plasma/whole blood concentration (T-max) | Up to day 17
Terminal elimination half-life (T-HALF) | Up to day 17
Apparent total body clearance (CL/F) | Up to day 17
Apparent volume of distribution of terminal phase (Vz/F) | Up to day 17
Percent of BMS-986322 plasma AUC(INF) relative to plasma radioactivity AUC(INF) (%AUC(INF)) | Up to day 17
Total radioactivity (TRA) ratio of blood AUC(INF) to plasma AUC(INF) | Up to day 17
Total amount of radioactivity recovered in urine (UR) | Up to day 17
Percent of total amount of radioactivity recovered in urine (%UR) | Up to day 17
Total amount of radioactivity recovered in feces (FR) | Up to day 17
Percent of total amount of radioactivity recovered in feces (%FR) | Up to day 17
Total amount of radioactivity recovered in urine and feces combined (RTotal) | Up to day 17
Percent of total amount of radioactivity recovered in all excreta (%Total) | Up to day 17

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to day 47
Number of participants with serious adverse events (SAEs) | Up to day 47
Number of participants with AEs leading to discontinuation | Up to day 47
Number of participants with vital sign abnormalities | Up to day 17
Number of participants with electrocardiogram (ECG) abnormalities | Up to day 17
Number of participants with clinically significant physical examination findings | Up to day 17
Number of participants with clinical laboratory abnormalities | Up to day 17

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Fortrea Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-andresearch/ disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html